CLINICAL TRIAL: NCT03191175
Title: Residual Immune Activation in HIV-infected Patients on Successful cART: Association Between Inflammasome Activation in Monocytes by Circulating Metabolites and Non AIDS Defining Comorbidities
Brief Title: Inflammasome Activation Via Circulating Metabolites
Acronym: InflammoVIH
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government); Sidaction (Other); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/14
Record Dates: First submitted 2017-06-14; First posted 2017-06-19 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Inflammasome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV patients
  Interventions: Other: blood sample
- Control patients
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — 47ml blood (40 ml EDTA whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation and 7 ml for serum).

SUMMARY:
The clinical challenges confronting patients with HIV has shifted over the past 10 years from acquired immunodeficiency syndrome to chronic diseases including atherosclerosis, neurocognitive disorders, and osteoporosis. Chronic low grade inflammation and monocyte activation have been consistently associated with comorbidities in HIV patients. Indeed, recent studies indicate that inflammatory mediators including IL-6, IL-1, sCD14 and s CD163 produced by monocytes, but not T-cell activation, predict Non-AIDS-related events in virologically suppressed HIV-infected persons treated with combined antiretroviral therapy (cART), highlighting the important role of monocyte activation in the occurrence of comorbidities in cART-treated HIV infected patients. Yet, the underlying molecular pathways of persistent monocyte activation in cART treated HIV-infected patients remains incompletely characterized. Our preliminary results: 1/ establish a link between the activation of the inflammasome, the increased of pyrimidine-derived metabolites and the cardiovascular risk in a cohort of elderly patients; 2/ show that treated HIV-patients are characterized by increased soluble IL-1b or IL-18 in their blood suggesting that the inflammasome pathway is activated.

Objectives: In this study we will characterize the molecular pathways underlying persistent monocyte activation in treated HIV patients, through the implication of the activation of the inflammasome machinery: 1. Characterization of NOD like Receptor (NLR) expression in monocytes for IL-1b and IL-18 secretion (inflammasome activation); 2. Characterization of circulating metabolites that active the inflammasome machinery; 3. Evaluation of the link between the activation of the inflammasome, the increased of circulating metabolites and the non-AIDS related comorbidities.

ELIGIBILITY:
HIV patients :

Inclusion Criteria:

* Aged 18 years and above
* HIV-1 infected patients
* Enrolled in the CIADIS substudy of the ANRS CO3 Aquitaine cohort
* Patients receiving antiretroviral therapy
* HIV-1 RNA load below the detection limit of 40 copies/mL
* With a written and signed informed consent

Exclusion Criteria:

* HIV-2 or HIV-1/HIV-2 co-infection

Control patients :

Inclusion Criteria:

* Aged 18 years and above

Exclusion Criteria:

* HIV-1, HIV-2 or HIV-1/HIV-2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients with long-term suppressed viral load on cART
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Characterization of NLR (s) implicated in IL-18 up-regulation (inflammasome activation) in HIV | At baseline (D0)
  * The metabolic profile in purified monocytes from HIV patients through label-free proteomics and assignment of metabolic targets
  * The expression of NLR genes by quantitative Polymerase Chain Reaction (qPCR) in purified monocytes from HIV patients.

SECONDARY OUTCOMES:
Characterization of circulating metabolites that active the inflammasome machinery | At baseline (D0)
  * analysis of the ability of sera from HIV patients to activate inflammasome in HIV negative monocytes, and to induce IL-1, IL-18, or both secretion.
  * metabolomic profile
  * analysis of the ability of predominant metabolites in HIV patients to activate inflammasome.
Non-AIDS related comorbidities | At baseline (D0)
  metabolites of interest, inflammasome activation measured by IL-1b and IL-18

CONTACTS AND LOCATIONS:
Overall Officials: Linda WITTKOP, MD, PhD, Study Chair — Université de Bordeaux - ISPED - Inserm 2129 - CHU de Bordeaux; Isabelle PELLEGRIN, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Benjamin FAUSTIN, PhD, Study Director — Centre National de la Recherche Scientifique, France
Locations (1):
- Service d'immunologie, Bordeaux, France

REFERENCES:
- [Background] Furman D, Chang J, Lartigue L, Bolen CR, Haddad F, Gaudilliere B, Ganio EA, Fragiadakis GK, Spitzer MH, Douchet I, Daburon S, Moreau JF, Nolan GP, Blanco P, Dechanet-Merville J, Dekker CL, Jojic V, Kuo CJ, Davis MM, Faustin B. Expression of specific inflammasome gene modules stratifies older individuals into two extreme clinical and immunological states. Nat Med. 2017 Feb;23(2):174-184. doi: 10.1038/nm.4267. Epub 2017 Jan 16. PMID 28092664
- [Background] Ozanne A, Duffau P, Dauchy FA, Rigothier C, Terrien C, Lazaro E, Cazanave C, Lawson-Ayayi S, Bonnet F, Blanco P, Wittkop L, Pellegrin I; CIADIS sub-study in the ANRS CO3 Aquitaine cohort study group. Activation, senescence and inflammation markers in HIV patients: association with renal function. AIDS. 2017 May 15;31(8):1119-1128. doi: 10.1097/QAD.0000000000001461. PMID 28328797
- [Background] Duffau P, Wittkop L, Lazaro E, le Marec F, Cognet C, Blanco P, Moreau JF, Dauchy FA, Cazanave C, Vandenhende MA, Bonnet F, Thiebaut R, Pellegrin I; ANRS CO3 Aquitaine Cohort Study Group. Association of immune-activation and senescence markers with non-AIDS-defining comorbidities in HIV-suppressed patients. AIDS. 2015 Oct 23;29(16):2099-108. doi: 10.1097/QAD.0000000000000807. PMID 26544576
- [Background] Wittkop L, Bitard J, Lazaro E, Neau D, Bonnet F, Mercie P, Dupon M, Hessamfar M, Ventura M, Malvy D, Dabis F, Pellegrin JL, Moreau JF, Thiebaut R, Pellegrin I; Groupe d'Epidemiologie Clinique du SIDA en Aquitaine. Effect of cytomegalovirus-induced immune response, self antigen-induced immune response, and microbial translocation on chronic immune activation in successfully treated HIV type 1-infected patients: the ANRS CO3 Aquitaine Cohort. J Infect Dis. 2013 Feb 15;207(4):622-7. doi: 10.1093/infdis/jis732. Epub 2012 Nov 29. PMID 23204178